CLINICAL TRIAL: NCT02049242
Title: Triple Tourniquet vs. Single Tourniquet at Open Myomectomy to Reduce Blood Loss: A Prospective Randomised Controlled Trials
Brief Title: Uterine Tourniquet at Open Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Erzurum Nenehatun Kadın Doğum Hastanesi (Unknown)
Responsible Party: Principal Investigator, Ragıp Atakan Al, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: atauni10
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Myomectomy; Uterine Leiomyoma
Keywords: Hemorrhage; Leiomyoma; Myofibroma; Uterine Myomectomy; Tourniquet
MeSH Terms: conditions — Myofibroma; Hemorrhage; Leiomyoma | interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple tourniquet (Active Comparator)
  Interventions: Procedure: triple tourniquet
- Single tourniquet (Active Comparator)
  Interventions: Procedure: Single tourniquet

INTERVENTIONS:
Procedure: triple tourniquet — Triple tourniquet consist of two tourniquet applied both infundibulopelvic ligaments and one uterine isthmus to occlude the left and right ovarian vessels and to occlude the uterine arteries. For this purpose, a small opening is made in the avascular place of the broad ligament on either side of the uterine isthmus superior to the uterine vessels. A pediatric Foley catheter is threaded through the two holes and tied tightly anteriorly around the cervix at the level of the internal os.
  Through the same openings in the broad ligament each side a Foley catheter looped around the infundibulopelvic ligament lateral to the fallopian tube and ovary.
  Arms: Triple tourniquet
Procedure: Single tourniquet — Single tourniquet is tourniquet applied uterine isthmus to occlude the uterine arteries. For this purpose, a small opening is made in the avascular place of the broad ligament on either side of the uterine isthmus superior to the uterine vessels. A pediatric Foley catheter is threaded through the two holes and tied tightly anteriorly around the cervix at the level of the internal os.
  Arms: Single tourniquet

SUMMARY:
The aim of study is to compare triple tourniquet vs. single tourniquet to reduce blood loss at open myomectomy.

DETAILED DESCRIPTION:
Single tourniquet is applied to uterine isthmus to occlude uterine arteries. Triple tourniquet is applied to both infundibulopelvic ligaments and uterine isthmus.

ELIGIBILITY:
Inclusion Criteria:

* uterine myoma >12 weeks

Exclusion Criteria:

* Pedunculated myoma, broad ligament myoma
* Hb<10.5 g /dl

Ages: 16 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Estimating blood loss at the end of myomectomy | 15 minutes postoperatifly
  Surgical blood loss will be estimated by sum of the volume of suction fluid and blood loss quantitated by gravimetric method.
  During surgery, if it is possible, irrigation will not be done, surgical sponge and compress will not be used.
  * Suction fluid will be measured at the end of operation and volume of irrigation fluid will be subtracted from total suction volume.
  * Surgical drapes, sponges and towels will be weighted before and just after surgery. The blood loss will be estimated as differences in gram by weighing when 1ml blood supposed as 1 gr.

SECONDARY OUTCOMES:
The amount of transfusions | 7 Days
  Erythrocyte transfusions transfusion will be allowed when haemoglobin dropped below 8 g/dL.
A change in hemoglobin | At baseline and 48 hours after surgery
Volume in drains | 7 days
  Drain will be removed when discharge drops below 50 ml/day
Anti-Mullerian Hormone levels variation | 6 weeks
  Anti-Mullerian Hormone levels before and 6 months after surgery

OTHER OUTCOMES:
Peri-operative complications | 6 weeks postoperatively
  Including but not limited to fever, pelvic infections, wound infections.
Total operation time | 5 minutes post operatively
Tourniquet time | 5 minutes after tourniquet removed

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Universitesi Araştırma Hastanesi, Erzurum, Yakutiye, Turkey (Türkiye)